CLINICAL TRIAL: NCT01651065
Title: Micro-Clinic Obesity and Metabolic Risk Prevention Program: A Randomized-Control Trial of a Social-Network Based Intervention
Brief Title: Micro-Clinic Obesity and Metabolic Risk Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microclinic International (Other)
Collaborators: Bell County Department of Health, Kentucky (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20110766
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type II; Heart Disease; Obesity; Hypertension; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases; Obesity; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microclinic Social Network Program (Experimental): Subjects will be receiving a 10/9-month Microclinic Diabetes Education Program (Team Up 4 Health) and 6 months of follow up. In the intervention these subjects will engage in the Microclinic Program support groups. The intervention program consists of 25 event sessions. Sessions are offered weekly the first month, and biweekly thereafter.
  Interventions: Behavioral: Microclinic Diabetes Education Program
- Active Controls (Active Comparator): Individuals will receive screening by clinical staff. Control group subjects are offered standard of care from local health department, but will not participate in program activities, other than offered option to join open-community health events.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Microclinic Diabetes Education Program — The microclinic intervention leverages different levels of social networks to positively influence behaviors relating to diabetes and other metabolic conditions through small treatment units called, 'microclinic groups (MC),' consisting of 2-6 friends and family members of the same social network, which lead to a larger network of 'classes' and cohorts.
  The program provides MC subjects with shared access to health education and group support to promote glycemic and metabolic control through diet, exercise, and treatment adherence. MC members play a role in the collective effort to combat diabetes and solidifying self-management behavioral skills through peer-monitoring and encouragement of lifestyle behaviors.
  Arms: Microclinic Social Network Program
Behavioral: Control
  Arms: Active Controls

SUMMARY:
The purpose of this randomized trial is to study the efficacy of a novel social propagation intervention which integrates social network induction with health education for weight and metabolic control among patients with type 2 diabetes, BMI of 25-30+, and cardiovascular disease. The intervention takes place in the form of a community health program, where participants who enroll in this program will be asked if they would like to take part in the study to evaluate its efficacy. Thus, the investigators will study the efficacy of social networks in propagating changes in lifestyle factors for diabetes and chronic disease management

DETAILED DESCRIPTION:
The potential to harness the propagating power of social networks for chronic disease treatment and management, such as for diabetes and obesity, is an emerging area in epidemiology and clinical research. Social induction for disease management has been effectively leveraged for disease management, but we have not carefully disaggregated of different layers and modalities of social network effects in this context. This study will test and demonstrate this through a novel randomized trial.

The randomized design is comprised of 2 arms. 1) Intervention Group: This arm takes part in a 10-month (9-month for Phase 2, cycles 1 and 2) diabetes, weight, and cardiovascular disease education and management program in combination with the microclinic social support model. A microclinic is a support group of 2-6 individuals from the same social network who learn how to manage their disease together. 2) Control Group: This is a control arm with observational parallel assessments of metabolic and lifestyle risk factors alone (implemented in Phase 1 and 2, cycles 1 and 2). Each arm will take part in a 6-month follow-up. The investigators also aim to study the intervention effects of social networks in improving lifestyle risk factors on a small sample of Phase 1 controls in a repeated measures design. Observational controls with 7 repeated measures in Phase 1 (pre-intervention) will receive the 9-month diabetes, weight, and cardiovascular disease education and management program with microclinic social support model condensed in a 4-6 months program. The controls in this cycle will also receive 17 medical screenings during the intervention, and 6-month follow-up (post-intervention).

Aim 1- (Phase 1 and 2, Cycles 1 & 2)

To evaluate the efficacy of the microclinic intervention group versus observational control in improving lifestyle factors and metabolic outcome.

Aim 2- (Phase 2, Cycle 3)

To examine the effect of the microclinic intervention by comparing pre- and post measures among those who were first controls in Phase 1 and then participated in the microclinic intervention Phase 2, Cycle 3.

AIM 3- (Phases 1 & 2, cycles 1, 2, and 3)

To differentiate the modalities of social network effects: direct causal induction versus homophilly, and to determine the extent of long-term temporal cross-propagating effects between-persons in a microclinic group.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in our community health program.
* Over the age of 18
* BMI of 30 or higher, or
* BMI of 25 or higher AND must be diagnosed with at least one additional risk factor 1) type 2 diabetes, 2) high blood pressure, and/or 3) high cholesterol
* For those who will be participating in the cross-over sub-sample, they must have previously participated in Phase 1 as subject of the control group, or

Exclusion Criteria:

* Patients who are not enrolled in the our community health education program (applies to Phase 1 only)
* Are not able to provide informed consent for themselves
* Under the age of 18
* Has undergone weight loss surgery
* Pregnant women*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Weight | From baseline until end of intervention period (9-10 months), and 6 months post-intervention
  Change in weight over time

SECONDARY OUTCOMES:
Waist circumference | From baseline until end of intervention period (9-10 months), and 6 months post-intervention
  Change in waist measurement over time
Blood pressure | From baseline until end of intervention period (9-10 months), and 6 months post-intervention
  Change in systolic/diastolic blood pressure over time
HDL | From baseline until end of intervention period (9-10 months), and 6 months post-intervention
  Change in HDL over time
Hemoglobin A1c (%, HbA1c) | From baseline until end of intervention period (9-10 months), and 6 months post-intervention
  Change in HbA1c over time

OTHER OUTCOMES:
Social network induction and clustering | From baseline to end of intervention period (9-10 months)
  Investigate the magnitude of social network-driven clustering (via hierarchal multilevel analysis) on the longitudinal trajectories of body mass, lipids, and HbA1c changes. Specifically, assess the relative magnitude of intraclass correlation of microclinics, classroom, cohort, and geographic neighborhoods.
Temporally investigate the causal induction of cascading changes in body weight between follow-ups on subsequent weight changes in other participants. | Change from each regularly scheduled classroom session, on each subsequent session, during intervention period.
  Using time intervals between follow-ups analyzed as separate induction timeframe windows, we estimate how weight loss observed in a previous time window predicts body weight change in subsequent followup intervals of the other participants.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Zoughbie, D.Phil., Principal Investigator — Microclinic International; Eric L Ding, Sc.D., Principal Investigator — New England Complex Systems Institute
Locations (1):
- Bell County Health Department, Pineville, Kentucky, United States

REFERENCES:
- [Derived] Ding EL, Watson KT, Makarechi L, James Ng TL, Huddleston D, Bui N, Tsai LL, Zoughbie DE. Social Induction via a Social Behavioral Intervention on Changes in Metabolic Risk Factors: A Randomized Controlled Trial in Rural Appalachia, United States. Mayo Clin Proc. 2024 Jul;99(7):1058-1077. doi: 10.1016/j.mayocp.2023.11.023. PMID 38960495
- See also: Related Info — http://microclinics.org